CLINICAL TRIAL: NCT06644092
Title: Investigation of the Effectiveness of Physiotherapy and Rehabilitation After Osteochondral Allograft Transplantation Operation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, YagmurOrta, Yeditepe University, Yeditepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YagmurOrta
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cartilage Damage; Osteochondral Lesion; Allograft; Osteoarthritis of Knee
Keywords: Physical Therapy; Osteochondral Allograft Transplantation; Osteochondral Lesion; Cartilage Damage
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigation of the Effectiveness of Physiotherapy and Rehabilitation After Osteochondral Allograft (Experimental): The question of our research is to determine the effectiveness of the physiotherapy and rehabilitation protocol applied in the postoperative period on the knee joint range of motion, functionality, muscle strength around the knee joint (quadriceps/hamstring ratio) and pain parameters in patients who underwent osteochondral allograft transplantation surgery and to include it in the literature. In this direction, the hypotheses of our study are; H0: The physical therapy and rehabilitation protocol to be applied after osteochondral allograft transplantation surgery has a positive contribution to the patient's knee joint range of motion, functionality, muscle strength and pain.
  H1: The physical therapy and rehabilitation protocol to be applied after osteochondral allograft transplantation surgery does not have a positive contribution to the patient's knee joint range of motion, functionality, muscle strength and pain.
  Interventions: Other: Investigation of the Effectiveness of Physiotherapy and Rehabilitation After Osteochondral Allograft Transplantation Operation

INTERVENTIONS:
Other: Investigation of the Effectiveness of Physiotherapy and Rehabilitation After Osteochondral Allograft Transplantation Operation — The treatment protocol to be applied to the patients after surgery was determined. The protocol includes; cold application, game ready device application, CPM device application, patellar mobilization, soft tissue mobilization application, TENS, conventional TENS and NMES application, ultrasound application, stretching exercises, strengthening exercises, mobilization exercises, balance and proprioception exercises, walking training and kinesio taping.

SUMMARY:
The aim of our study is to add to the literature the effect of the effectiveness of the physiotherapy and rehabilitation in the clinic, which will be applied to the patients after the osteochondral allograft transplantation operation, which is a current treatment approach applied after knee cartilage tissue damage, on the range of motion, functionality, pain and muscle strength of the patients during the recovery process. The clinical importance of our aim is that it will have the potential to guide health professionals in determining the appropriate treatment approach in order to reveal the best results that can be obtained due to the lack of many studies in the literature on the treatment of patients after osteochondral allograft surgery.

ELIGIBILITY:
Inclusion criteria:

Patients who underwent osteochondral allograft transplantation surgery Participant's acceptance/desire to participate in the study

Exclusion criteria:

Patient participant's refusal/desire to participate in the study Inability to perform exercises due to infection etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-04-09 (Estimated); Study Completion 2025-05-09 (Estimated)

PRIMARY OUTCOMES:
KOOS | 6 months
  Knee Injury and Osteoarthritis Outcome Score (KOOS): A health measure used to evaluate knee injuries and knee-related conditions such as osteoarthritis. The KOOS comes in a widely used questionnaire format to assess patients' knee function, pain, quality of life, and other symptoms. By measuring problems in subcategories such as pain, symptoms, quality of life, functional limitations, and sports/dialysis activities, it provides healthcare professionals with an important tool to monitor patients' response to treatment, evaluate treatment plans, and understand patients' quality of life.
Oxford Knee Scale | 6 months
  The Oxford Knee Score (ODS) is a valid and reliable questionnaire with a Turkish version that allows individuals with knee OA to assess their own function and pain. It is scored on a Likert scale from 0 (absent) to 4 (severe) (0-48). In this questionnaire consisting of 12 questions, questions 2, 3, 7, 11 and 12 assess functional status; questions 1, 4, 5, 6, 8, 9 and 10 assess pain-related status. Scores from ODS pain questions range from 0 to 28 points, with the lowest score being 0 and the highest score being 28. Scores from ODS function 30 parameters range from 0 to 20 points, with the lowest score being 0 and the highest score being 20. High scores indicate worse functional status and pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe University Hospital, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Nho SJ, Pensak MJ, Seigerman DA, Cole BJ. Rehabilitation after autologous chondrocyte implantation in athletes. Clinics in sports medicine. 2010 Apr 1;29(2):267-82. 2. Flanigan DC, Harris JD, Trinh TQ, Siston RA, Brophy RH. Prevalence of chondral defects in athletes' knees: a systematic review. Med Sci Sports Exerc. 2010 Oct 1;42(10):1795-801. 3. Moyad TF. Cartilage injuries in the adult knee: evaluation and management. Cartilage. 2011 Jul;2(3):226-36. 4. Hjelle K, Solheim E, Strand T, Muri R, Brittberg M. Articular cartilage defects in 1,000 knee arthroscopies. Arthroscopy: The Journal of Arthroscopic & Related Surgery. 2002 Sep 1;18(7):730-4. 5. Chimutengwende-Gordon M, Donaldson J, Bentley G. Current solutions for the treatment of chronic articular cartilage defects in the knee. EFORT open reviews. 2020 Mar 2;5(3):156-63. 6. Berta Á, Duska Z, Tóth F, Hangody L. Clinical experiences with cartilage repair techniques: outcomes, indications, contraindications and rehabilitation. Joint Diseases and Related Surgery. 2015;26(2):084-96. 7. Cole BJ, Haunschild ED, Carter T, Meyer J, Fortier LA, Gilat R, ... & Pace JL. Clinically significant outcomes following the treatment of focal cartilage defects of the knee with microfracture augmentation using cartilage allograft extracellular matrix: a multicenter prospective study. Arthroscopy: The Journal of Arthroscopic & Related Surgery. 2021 May;37(5):1512-1521. 8. Vogt S, Angele P, Arnold M, Brehme K, Cotic M, Haasper C, Hinterwimmer S, Imhoff AB, Petersen W, Salzmann G, Steinwachs M. Practice in rehabilitation after cartilage therapy: an expert survey. Archives of orthopaedic and trauma surgery. 2013 Mar;133:311-20. 9. Krych AJ, Saris DB, Stuart MJ, Hacken B. Cartilage injury in the knee: assessment and treatment options. JAAOS-Journal of the American Academy of Orthopaedic Surgeons. 2020 Nov;28(22):914-922. 10. Crowley SG, Pedersen A, Fortney TA, Swindell HW, Saltzman BM, Popkin CA, Trofa DP. Rehabilitation variability fo